CLINICAL TRIAL: NCT07113041
Title: Neuromodulation-Enhanced Use of RObotic BALANCE Training to Improve Balance Function in Individuals With Stroke
Acronym: NEUROBALANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Vikram Shenoy Handiru, Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-1279-24; 90REGE0025-01-00 (Other Grant/Funding Number: National Institute for Disability, Independent Living, and Rehabilitation Research (NIDILRR))
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Stroke (CVA) or Transient Ischemic Attack; Stroke Ischemic; Stroke Gait Rehabilitation; Balance Deficits
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The mode of HD-tDCS (active/sham) will be masked for the participant, the study investigator, and the outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- RBT + Active HD-tDCS Group (Experimental): Participants will engage in balance and postural control training on a robotic balance platform called Hunova (Movendo, Italy). Before balance training, the current intensity of 2 mA will be delivered to the leg motor area identified using individual MRI-guided neuronavigated transcranial magnetic stimulation (nTMS), and the stimulation will be turned ON for 20 minutes.
  Interventions: Device: Combined (Robotic balance training and high-definition transcranial direct current stimulation)
- RBT + Sham HD-tDCS Group (Sham Comparator): Participants will engage in balance and postural control training on a robotic balance platform called Hunova (Movendo, Italy). Before balance training, the current intensity of 2 mA will be delivered to the leg motor area identified using individual MRI-guided neuronavigated transcranial magnetic stimulation (nTMS), and the stimulation will be turned ON transiently for 30 s to provide a sensation of stimulation.
  Interventions: Device: Combined (Robotic balance training and high-definition transcranial direct current stimulation)
- SOC Control Group (Other): The standard of care (SOC) control group participants will perform dose-matched conventional physical therapy exercises delivered by a trained PT.
  Interventions: Other: Standard of Care Balance Training

INTERVENTIONS:
Device: Combined (Robotic balance training and high-definition transcranial direct current stimulation) — The robotic platform will train the participants to maintain dynamic balance in the sagittal and transverse planes (mediolateral and anterior-posterior directions) and engage in core stability and trunk control with seated balance exercises. In addition, high-definition transcranial direct current stimulation (HD-tDCS) will be used as an adjuvant to robotic balance training by priming the corticospinal circuits.
  Arms: RBT + Active HD-tDCS Group; RBT + Sham HD-tDCS Group
Other: Standard of Care Balance Training — Participants in this group will receive a standard-of-care balance training (dose matched to the experimental group) administered by the Physical therapist.
  Arms: SOC Control Group

SUMMARY:
Our proposed study, "NEUROBALANCE Stroke,"; aims to evaluate the effectiveness of a combined intervention involving robotic balance training and noninvasive brain stimulation in improving balance function and postural control in individuals with chronic stroke. The study will recruit 45 participants who have had a stroke at least 6 months before enrolment and experience persistent balance and gait deficits. Participants will be randomized into three groups: (1) robotic balance training with active brain stimulation, (2) robotic balance training with sham brain stimulation, and (3) standard-of-care rehabilitation.

The study will involve 15 training sessions over 5 weeks, with assessments conducted at baseline, post-training, and two months post-training to evaluate balance recovery and retention. The primary focus is understanding how this intervention affects brain and muscle activity during balance tasks and how these changes translate into functional improvements in clinical outcome measures of balance function. Additionally, participant feedback on brain stimulation and exercise engagement will be collected to inform future studies.

The findings may guide the development of personalized training protocols and contribute to broader rehabilitation strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18-75 years
2. Diagnosed with a cortical/subcortical ischemic stroke at least 6 months before the screening, as confirmed by the neurological exam or an MRI.
3. Have complaints of impaired balance and poor postural control determined by a BBS score of ≤50.
4. Ability to stand upright with or without support for at least 20 seconds
5. Ability to walk with or without a walking aid for at least ten meters
6. Not planning to change medication in the next four months
7. Minimum Cognitive Ability to understand the verbal instructions and comply with the study procedures, as determined by the University of California, San Diego, Brief Assessment of Capacity to Consent Instrument (UBACC).

Exclusion Criteria:

1. Currently undergoing any regular physical therapy program or research studies focusing on balance functions.
2. Having a brainstem stroke.
3. Contraindication for MRI scan (presence of metal implants, claustrophobia)
4. Affected by the peripheral nerve injury, neuromuscular conditions, or orthopedic issues of lower limbs before stroke, or have any persistent pain or difficulty maintaining blood pressure while upright.
5. Have a scalp or skin condition (e.g., psoriasis or eczema) * on the scalp near the stimulation site
6. Having severe visual impairment (e.g., spatial neglect) or hearing problems that may affect study compliance
7. Any other neurological injury or psychiatric conditions (e.g., severe anxiety or schizophrenia etc.)
8. Contraindications to MRI, including the presence of non-titanium metallic implants, claustrophobia, etc.
9. Not be pregnant or thinking of becoming pregnant
10. Diagnosed with alcohol or substance abuse in the last 3 years
11. Contraindications to TMS, including the presence of metallic implants in the head and a history of seizures or medication-resistant epilepsy or ongoing use of anti-seizure/seizure threshold-lowering medications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | Baseline, post 5-week training, 2-month follow-up
  A widely used outcome measure of static standing balance function (Newstead et al., 2005), categorized under the 'Activity' subsection of ICF domain. BBS scores range from 0 to 56 (the higher, the better). The change in BBS scores from baseline to 4 weeks post-training will be the primary endpoint.

SECONDARY OUTCOMES:
Functional Gait Assessment (FGA) | Baseline, post 5-week training, and 2-month follow-up
  To assess dynamic balance during walking, unlike BBS, it is not prone to the ceiling effect(Van Bloemendaal et al., 2019). FGA will be used as the secondary outcome measure of balance function and gait. FGA comes under the ICF domains of 'Activity' and 'Body Function.'
Mini Balance Evaluation Systems Test (MBT) | Baseline, post 5-week training, and 2-month follow-up
  To identify the risk of falls (Yingyongyudha et al., 2016) with a high internal consistency with BBS and similar advantage of FGA, i.e., no ceiling effect. MBT will be used as the secondary endpoint of the balance function.
Trunk Impairment Scale (TIS) | Baseline, post 5-week training, and 2-month follow-up
  To estimate the trunk motor impairment(Verheyden et al., 2004). The scale ranges from 0 to 23 and assesses static and dynamic postural control.
Center of Pressure (COP) Displacement | Baseline, post 5-week training, and 2-month follow-up
  To evaluate the body sway in response to the perturbations of the posturography platform.
TMS-evoked EEG Potentials (TEP) | Baseline, post 5-week training, and 2-month follow-up
  A neurophysiological outcome measure of cortical reactivity. TEPs can directly measure cortical reactivity without being affected by the distal components of the nervous system, especially in neurological populations(Keser et al., 2022). In contrast to motor-evoked potentials, TEPs also offer the advantage of eliciting cortical responses at TMS intensity below the resting motor threshold.
EEG Corticocortical Functional Connectivity | Baseline, post 5-week training, and 2-month follow-up
  The imaginary part of coherence (iCOH) measured from the source-space EEG time-series will be used as an outcome measure of corticocortical connectivity, representing sensorimotor functional integration.
EEG-to-EMG Corticomuscular Connectivity | Baseline, post 5-week training, and 2-month follow-up.
  EG-to-EMG directed transfer function (DTF) will be used as an outcome measure of causal information flow from cortical areas to the leg muscles (Artoni et al., 2017; Peterson and Ferris, 2019). This measure is intended to capture changes in the efferent communication due to combined interventions.
EMG Muscle Coactivation | Baseline, post 5-week training, and 2-month follow-up.
  EMG co-contraction index will be used as an outcome measure of muscle activation between the antagonist and agonist muscle pair involved in reactive balance control.
Diffusion Tensor Imaging (DTI) Fractional Anisotropy | Baseline and post-5-week training
  The intervention-related changes in the structural neuroplasticity will be measured using the baseline-to-post-5-week-training changes in the Fractional Anisotropy Laterality Index (FALI) computed from the bilateral corticospinal tracts.

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Shenoy Handiru,, PhD, Principal Investigator — Kessler Foundation; Guang Yue, PhD, Study Director — Kessler Foundation; Gail Forrest, PhD, Study Director — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
We will submit the IPD available in the tabular data to the ICPSR after removing any personal or private identifiers. The neuroimaging and neurophysiological data (such as the MRI, EEG, TMS, and EMG) will be shared on OpenNeuro.org (or a similar platform) in a BIDS-standardized format.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Six months after study completion.
Access Criteria: "Authorized Users" (i.e., all Users with an account on the ICSPR) will have access to the data.
URL: https://www.icpsr.umich.edu/web/pages/index.html